CLINICAL TRIAL: NCT02670876
Title: Effectiveness of an Anti-bullying Intervention for Adolescent Perpetrators: Using Tools Measuring Brain Function and Structure, Cognition and Behavior.
Brief Title: Effectiveness of an Anti-bullying Intervention for Adolescent Perpetrators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Childrens Hospital (Other)
Responsible Party: Principal Investigator, Booog Nyung Kim, Professor, Seoul National University Childrens Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0720152106
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Conduct Disorder
MeSH Terms: conditions — Conduct Disorder

ARMS (1):
- Anti-bullying intervention (Experimental): An anti-bullying intervention target to perpetrators of school bullying was conducted. The program consisted of 8 sessions over 4 weeks and was conducted by a board-certified psychiatrist and a therapist with previous training in psychosocial treatments. The intervention was based on cognitive-behavioral therapy (CBT) principles and addressed various factors that have been associated with perpetrators of school bullying, including impulse control, perspective taking (empathy), and the enhancement of communication skills.
  Interventions: Behavioral: Anti-bullying intervention

INTERVENTIONS:
Behavioral: Anti-bullying intervention — The title of each session were as follows :
  1. Introduction of intervention and setting rules, building rapport
  2. Understanding school bullying (The definition of school bullying and proper coping strategies)
  3. Empathy of others ( Practice of understanding victims of school bullying)
  4. Impulse control 1 (Understanding my anger patterns, finding one's true feelings behind that anger)
  5. Impulse control 2 (Finding irrational thoughts that lead to anger and correction of them)
  6. Conflict management (Understanding one's pattern of dealing with conflicts, finding effective strategies)
  7. Communication skills enhancement
  8. Increasing self esteem

SUMMARY:
The investigators recruited school bullying perpetrators from the age of 12 to 17 by referral from the local police department. An anti-bullying intervention based on cognitive-behavioral therapy (CBT) principles was conducted, and addressed issues related to impulse control, empathy and communication enhancement. All participants completed brain magnetic resonance imaging, neurocognitive tests, and questionnaires before and after the intervention.

DETAILED DESCRIPTION:
The present study included previous perpetrators of school bullying who were convicted for a minor offense, including physical or verbal assaults or theft, and who were referred by the police to participate in an anti-bullying intervention. The program consisted of 8 sessions over 4 weeks and was conducted by a board-certified psychiatrist and a therapist with previous training in psychosocial treatments. The intervention was based on CBT principles and addressed various factors that have been associated with perpetrators of school bullying, including impulse control, perspective taking (empathy), and the enhancement of communication skills.

All participants completed the Korean Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-PL) administered by board-certified child and adolescent psychiatrists. The validity and reliability of the original and Korean versions of the K-SADS-PL have been established. Intelligence quotient (IQ) was measured using the Korean Educational Developmental Institute's Wechsler Intelligence Scale for Children.

Prior to and after participation in the program, all participants underwent brain magnetic resonance imaging (structural and functional) and completed neurocognitive tests that included the continuous performance test (CPT), the Stroop Word and Color Test, and the Wisconsin Card Sorting Test (WCST). The parents of the participants completed questionnaires including the Child Behavior Checklist (CBCL). Written informed consent was obtained from the parents and the participants after sufficient explanation of the study. The study protocol was approved by the institutional review board of the Seoul National University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* No psychiatric diagnosis or psychiatric diagnoses including conduct disorder, depressive disorder, oppositional defiant disorder, attention-deficit hyperactivity disorder, and adjustment disorder.
* IQ > 70
* Agreement to participate
* Ability to cooperate in group therapy

Exclusion Criteria:

* Any psychotic disorder
* Severe impairment in impulse control
* Not cooperating with program participation
* IQ < 70
* Current or past history of brain trauma or organic brain disorder, seizure disorder, or any neurological disorder.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Brain activity measured by functional magnetic resonance imaging (fMRI) | 1 month

SECONDARY OUTCOMES:
Aggression measured by the Child Behavior Checklist based on parent-report | 1 month
Cognitive flexibility measured by the Wisconsin Card Sorting Test | 1 month

REFERENCES:
- [Derived] Kim JI, Kang YH, Lee JM, Cha J, Park YH, Kweon KJ, Kim BN. Resting-state functional magnetic resonance imaging investigation of the neural correlates of cognitive-behavioral therapy for externalizing behavior problems in adolescent bullies. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Aug 30;86:193-202. doi: 10.1016/j.pnpbp.2018.05.024. Epub 2018 Jun 6. PMID 29885469